CLINICAL TRIAL: NCT06040983
Title: Monocenter, Open Label Clinical Investigation on the Treatment of Radiation Induced Dermatitis With FR-101 Chest Dressing
Brief Title: Clinical Investigation on the Treatment of Radiation Induced Dermatitis With FR-101 Chest Dressing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chih-Ying Liao, Attending physician, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH112-REC1-001
Record Dates: First submitted 2023-09-01; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Radiation Dermatitis
Keywords: radiation-irritated skin
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FR-101 Dressing use (Experimental): Subject will use FR-101 chest dressing on the target skin area accepted radiation therapy once every 2 days.
  Interventions: Device: FR-101 Chest Dressing

INTERVENTIONS:
Device: FR-101 Chest Dressing — Subject will receive FR-101 chest dressing and be instructed to use the product on the target skin area accepted radiation therapy once every 2 days, taking care of avoiding applications from 1 to 4 h before treatment to prevent "Build-up" effect. If the application time is longer than the recommendation, discomfort may happen depending on subject's condition.

SUMMARY:
Breast cancer is the top one incidence of cancer in women. Whole breast radiation therapy plays an indispensable role in the course of breast cancer treatment, and the radiation dermatitis is the major side effect affected quality of life. Radiation dermatitis can be divided into acute and chronic. Severe acute radiation dermatitis affects the quality of life of patients during the course of treatment, and may cause treatment interruption and affect the efficacy. Chronic radiation dermatitis may cause irreversible skin problems, and lead to so-called "radiation-irritated skin" (radiation-irritated skin) seriously affects the quality of life of breast cancer patients after treatment.

This study will enroll 30 breast cancer patients who received whole breast radiation therapy after breast conserving surgery. Subject will receive FR-101 chest dressing and be instructed to use the product on the target skin area accepted radiation therapy once every 2 days, taking care of avoiding applications from 1 to 4 h before treatment to prevent "Build-up" effect.

Subjects will need to come back to clinics for assessment weekly during radiotherapy, 2 weeks after radiotherapy, and 6 weeks after radiotherapy. The evaluation includes physical examinations, questionnaire surveys, skin observation and measurements, and photographs. The total study time is at least 3 months. The target area of radiation-irritated skin condition will be observed and graded according to CTCAE rate. The skin physiological parameters will be detected by MoistureMeter SC, Vapometer, SkinColorCatch and HX-YL001 infrared thermometer.

Statistical analysis of skin physiological parameters is used to evaluate the efficacy of FR-101 chest dressing on the prevention of acute radiation dermatitis after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be males or non-pregnant females at least 20 years of age.
* Diagnosis of non-inflammatory breast adenocarcinoma or in situ breast cancer which were treated by operation with or without adjuvant or neoadjuvant hormonal treatment.
* Patients were scheduled to receive five sessions of radiotherapy per week (1 session per day) for at least four weeks using standard irradiation fraction (with at least 1.8 Gy per session) for total dose of at least 45 Gy or hypofraction irradiation fraction(with 2.66 Gy per session) for total dose of at least 42.56 Gy.
* Participant must give informed consent.

Exclusion Criteria:

* Bilateral breast cancer
* Previous radiotherapy to the chest
* Chemotherapy concurrent with radiation treatment
* Prior breast reconstructions, implants, and/or expanders
* Known radiosensitivity syndromes (e.g. Ataxia-telangiectasia)
* Collagen vascular disease, vasculitis, unhealed surgical sites, breast infections or systemic lupus erythematosus (SLE)
* Participation in any clinical trial in the prior 30 days from baseline.
* Any condition that, in the judgement of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-18 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Worst skin toxicity during treatment and until 2 weeks after according to CTCAE grading. | 1-Week (Day0), 2-Week (Day7), 3-Week (Day14), 4-Week (Day21), 5-Week (Day28), 6-Week (Day35), Post-radiotherapy 2 Week later
  Skin toxicity at the radiotherapy site will be assessed by investigator and NCI CTCAE v5.0 will be used for grading, on a scale of:
  Grade 1 (faint erythema or dry desquamation);
  Grade 2 (moderate to brisk erythema;patchy moist desquamation,mostly confined to skin foldsand creases; moderate edema);
  Grade 3 (moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion);
  Grade 4 (life-threatening consequences; skin necrosis or ulceration of full thickness dermis; spontaneous bleeding from involved site; skin graft indicated);
  Grade 5 (death)

SECONDARY OUTCOMES:
To compare the skin moisture percentage. | 1-Week (Day0), 3-Week (Day14), 5-Week (Day28), 6-Week (Day35), Post-radiotherapy 2 Week later, Post-radiotherapy 6 Week later
  To compare the skin moisture percentage at the radiotherapy site and normal site from baseline to follow-up visit.
To compare the skin trans-epidermal water loss. | 1-Week (Day0), Post-radiotherapy 2 Week later, Post-radiotherapy 6 Week later
  To compare the skin trans-epidermal water loss at the radiotherapy site and normal site from baseline to follow-up visit.
To compare the skin temperature of target region. | 1-Week (Day0), 3-Week (Day14), 5-Week (Day28), 6-Week (Day35), Post-radiotherapy 2 Week later, Post-radiotherapy 6 Week later
  To compare the skin temperature of target region at the radiotherapy site and normal site from baseline to follow-up visit.
The score of quality of life with the Skindex-16 questionnaire. | 1-Week (Day0), 3-Week (Day14), 5-Week (Day28), 6-Week (Day35), Post-radiotherapy 2 Week later, Post-radiotherapy 6 Week later
  The score of quality of life will be assessed using the Skindex-16 questionnaire every two weeks. Participants answer 16 questions on a scale from 0 (not at all) to 6 (always). The quality of life is calculated by summing the scores for all questions, resulting in a maximum of 96 and a minimum of 0; higher scores indicate a more impaired quality of life.
Median time to G2 radiation dermatitis development | 1-Week (Day0), 2-Week (Day7), 3-Week (Day14), 4-Week (Day21), 5-Week (Day28), 6-Week (Day35), Post-radiotherapy 2 Week later, Post-radiotherapy 6 Week later
  Median time to G2 radiation dermatitis development according to CTCAE.